CLINICAL TRIAL: NCT05566847
Title: Overcoming Therapeutic Inertia Among Adults Recently Diagnosed With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-21-OTI-02
Record Dates: First submitted 2022-09-21; First posted 2022-10-04 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Usual Care (No Intervention): Participants will receive standard care for newly diagnosed Type 2 Diabetes.
- Arm 2: Physician Education (Experimental): Physicians in service areas randomized to this arm were invited to a physician education session on therapeutic inertia.
  Interventions: Other: Physician Education
- Arm 3: Physician Education + Accountable Population Manager Outreach (Experimental): Physicians in service areas randomized to this arm were invited to a physician education session on therapeutic inertia. Patients enrolled in this arm may receive proactive outreach from an Accountable Population Manager (APM).
  Interventions: Other: Physician Education; Other: Accountable Population Manager outreach

INTERVENTIONS:
Other: Physician Education — The physician education session delivered to primary care physicians in Arms 2 and 3 will provide an educational update from the regional clinical leader for diabetes regarding guidelines for diabetes treatment and addressing therapeutic inertia.
  Arms: Arm 2: Physician Education; Arm 3: Physician Education + Accountable Population Manager Outreach
Other: Accountable Population Manager outreach — Patients will be referred to an Accountable Population Manager (APM) for proactive outreach, including supporting medication adherence and educational and overall support for T2D management. An APM is a non-physician clinician (for example, a clinical pharmacist) supporting diabetes management.
  Arms: Arm 3: Physician Education + Accountable Population Manager Outreach

SUMMARY:
Therapeutic inertia may result from providers, patients, and/or systems, but can be detrimental to a patients' health by putting them at risk for diabetes complications, though addressing it early can mitigate some of its effects. In Type 2 diabetes (T2D) care, this may look like failure to initiate metformin therapy early in the disease course. This project aims to evaluate the effects of proactive outreach by a non-physician clinician (Accountable Population Manager [APM]) to patients with newly diagnosed Type 2 diabetes. The team hypothesizes individuals receiving proactive outreach by an APM will be more likely to achieve glycemic targets at 6 months following start of the intervention.

DETAILED DESCRIPTION:
This is a 3-arm randomized clinical trial comparing patients in the following arms: 1) usual Type 2 diabetes care, 2) primary care physicians have been exposed to physician education on therapeutic inertia, and 3) primary care physicians have been exposed to physician education on therapeutic inertia and patients are referred to APM proactive outreach. The APM is a non-physician clinician, including clinical pharmacists and nurses. Eligible members will be identified via electronic health record (EHR) data in two stages: 1) identification of individuals with newly diagnosed T2D, 2) identification of the subset of newly diagnosed individuals with metformin-related therapeutic inertia. The content of the APM visit will be the same as what currently occurs in standard diabetes care, including discussing the risks and benefits of pharmacologic treatment and initiating treatment (with patient agreement), supporting medication adherence, and providing education and support for overall T2D management. The main outcome will be HbA1c at 6, 12, and 18 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Northern California (KPNC) member age 18-74
* Incident Type 2 Diabetes
* Patient of primary care physician (PCP) working in the randomized service areas
* Identified metformin-related therapeutic inertia
* At least one A1c 6.5-7.9 from 4 months post-diagnosis up to the time of randomization

Exclusion Criteria:

* Evidence of preceding T2D diagnosis
* Pregnant at the time of T2D diagnosis
* Likely to have Type 1 diabetes

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 817 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c<7% | 6 months
  Proportion of patients with HbA1c less than 7% at 6 months following the start of the intervention.
HbA1c<7% | 12 months
  Proportion of patients with HbA1c less than 7% at 12 months following the start of the intervention.
HbA1c<7% | 18 months
  Proportion of patients with HbA1c less than 7% at 18 months following the start of the .intervention.
HbA1c<8% | 6 months
  Proportion of patients with HbA1c less than 8% at 6 months following the start of the intervention.
HbA1c<8% | 12 months
  Proportion of patients with HbA1c less than 8% at 12 months following the start of the intervention.
HbA1c<8% | 18 months
  Proportion of patients with HbA1c less than 8% at 18 months following the start of the intervention.
HbA1c<9% | 6 months
  Proportion of patients with HbA1c less than 9% at 6 months following the start of the intervention.
HbA1c<9% | 12 months
  Proportion of patients with HbA1c less than 9% at 12 months following the start of the intervention.
HbA1c<9% | 18 months
  Proportion of patients with HbA1c less than 9% at 18 months following the start of the intervention.

SECONDARY OUTCOMES:
Time to achievement of glycemic targets (HbA1c<7%, <8%, and <9%) | 18 months
  Time elapsed
Adherence to HbA1c monitoring | 6 months
  New HbA1c value at follow-up time points
Adherence to HbA1c monitoring | 12 months
  New HbA1c value at follow-up time points
Adherence to HbA1c monitoring | 18 months
  New HbA1c value at follow-up time points
Time to metformin initiation | 18 months
  Time elapsed
Metformin adherence | 6 months
  Among those initiated on metformin, adherence to medication (proportion days covered, ≥80% vs. <80%)
Metformin adherence | 12 months
  Among those initiated on metformin, adherence to medication (proportion days covered, ≥80% vs. <80%)
Metformin adherence | 18 months
  Among those initiated on metformin, adherence to medication (proportion days covered, ≥80% vs. <80%)
Time to initiation of non-metformin anti-diabetes medication | 18 months
  Time elapsed
Absolute mean reduction in HbA1c from baseline | 6 months
  Absolute mean reduction in HbA1c from baseline to 6 months following intervention
Absolute mean reduction in HbA1c from baseline | 12 months
  Absolute mean reduction in HbA1c from baseline to 12 months following intervention
Absolute mean reduction in HbA1c from baseline | 18 months
  Absolute mean reduction in HbA1c from baseline to 18 months following intervention
Emergency room visits and hospitalizations post-intervention start | 18 months
  Emergency room visits and hospitalizations within 18 months of intervention start
Hypoglycemia events post-intervention start | 18 months
  Hypoglycemia events within 18 months of intervention start

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Gilliam, MD, PhD, Principal Investigator — Kaiser Permanente; Anjali Gopalan, MD, MS, Principal Investigator — Kaiser Permanente; Richard Grant, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Division of Research, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT05566847/Prot_000.pdf